CLINICAL TRIAL: NCT06488417
Title: Evaluation of Frankincense Essential Oil Supplements on Markers of Inflammation and Cellular Health
Brief Title: Frankincense Supplements and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dōTERRA International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DO-124033-FRA
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Frankincense essential oil; Boswellic acid; Gene expression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frankincense essential oil + boswellic acid supplement (Experimental): Participants in this arm take two capsules of a frankincense essential oil + boswellic acid supplement daily for approximately 30 days.
  Interventions: Dietary Supplement: Frankincense essential oil + boswellic acid supplement
- Frankincense essential oil supplement (Active Comparator): Participants in this arm take two capsules of a frankincense essential oil supplement daily for approximately 30 days.
  Interventions: Dietary Supplement: Frankincense essential oil supplement

INTERVENTIONS:
Dietary Supplement: Frankincense essential oil + boswellic acid supplement — This supplement contains frankincense essential oil and boswellic acid as its active ingredients.
  Arms: Frankincense essential oil + boswellic acid supplement
Dietary Supplement: Frankincense essential oil supplement — This supplement contains frankincense essential oil as its active ingredient.
  Arms: Frankincense essential oil supplement

SUMMARY:
The goal of this clinical trial is to learn whether frankincense essential oil-based supplements can affect gene expression and serum protein markers in healthy volunteers. The main questions it aims to answer are:

1. Do frankincense essential oil supplements affect gene expression and protein markers as measured in blood?
2. How does daily ingestion of frankincense supplements affect anthropometric measurements, including body mass index, waist circumference, blood pressure, and heart rate?
3. How does daily ingestion of frankincense essential oil supplements affect subjective quality of life and health parameters?
4. Is ingesting frankincense essential oil supplements daily safe, as measured by laboratory tests and adverse events?

Researchers will compare two types of frankincense essential oil supplements. One type contains frankincense essential oil and boswellic acid as its active ingredients. The other type contains only frankincense essential oil as its active ingredient.

Participants will:

* Be assigned one of the two types of frankincense essential oil supplement
* Take two capsules of their assigned supplement every day for about 30 days
* Attend two study visits in which they provide blood and urine samples, complete subjective health and quality of life assessments, and undergo anthropometric measurements
* Complete weekly subjective health assessments from home

DETAILED DESCRIPTION:
This randomized, double-blind study will recruit healthy men and women to compare gene expression profile and serum protein markers before and after consumption of frankincense essential oil supplements for approximately 4 weeks. Quality of life will also be assessed using subjective surveys and questionnaires. Safety markers (liver and kidney function, hematology, urinalysis, and adverse events) will be collected.

ELIGIBILITY:
Inclusion Criteria:

Males and females, 18-64 years old

* Willing to wash out of all internally-consumed essential oil and botanical products for at least 2 weeks prior to starting the study and willing to maintain the washout for the duration of the study (about 7 weeks)
* Local to Pleasant Grove, Utah, and/or willing to come to the clinical research center for study visits
* Willing to provide blood and urine samples during study visits
* Willing and able to consume study product daily for about 4 weeks
* Willing to track consumption of study product
* Willing to keep diet, exercise, sleeping, and current non-study supplement use the same throughout the study
* Willing to avoid alcohol, recreational drugs, and smoking/vaping for the duration of the study (approximately 5 weeks)
* Willing to wash out of internally-consumed essential oil and botanical products for approximately 7 weeks
* Willing to receive and respond to regular texts, emails, and/or phone calls from study staff
* No metabolic disease (BMI>35, diagnosis and treatment of hypertension, diabetes, or dyslipidemia)
* No major diseases under treatment by doctor (Medical Reviewer's discretion)
* No pregnancy within the last 60 days or currently breastfeeding (females)
* No allergy to olive oil, frankincense essential oil, or boswellic acid
* No internal consumption of frankincense oil regularly within the last 1 month (regularly is defined as dosing daily for more than 2 consecutive weeks, or dosing more than 2-3 times per week for 4 consecutive weeks)
* No alcohol, recreational drug, or smoking/vaping use in the past 1 month
* No evidence of medical condition, significant disease or disorder, medication, or surgery within the past 12 months that may, in the judgment of the medical provider, put the participant at risk or affect study results, procedures, or outcomes
* Not currently or previously participating in any other clinical trial within the last 30 calendar days
* Signed informed consent, HIPAA Authorization, and Confidentiality Agreement

Exclusion Criteria:

* Failure to meet any of the above inclusion criteria

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Gene expression | 4 weeks
  Gene expression analysis refers to a genome-wide quantification of methylation. EPIC850k array will be used for methylation analysis. This represents approximately 900,000 gene locations. The main feature performed is a differential methylation analysis to determine what has significantly changed from one time point to another.
Interleukin 6 (pg/mL) | 4 weeks
  Serum marker for inflammation
Fasting insulin (uIU/mL) | 4 weeks
  Serum marker used to determine whether insulin levels are affected by the consumption of the study product.
Matrix metalloproteinase-9 (ELISA) | 4 weeks
  Serum protein involved in inflammatory response and tissue remodeling
High sensitivity C-reactive protein (mg/L) | 4 weeks
  Serum marker for inflammation and cardiac health

SECONDARY OUTCOMES:
Albumin (g/dL) | 4 weeks
  Item in comprehensive metabolic panel for safety assessment
Blood urea nitrogen (BUN) (mg/dL) | 4 weeks
  Item in comprehensive metabolic panel for safety assessment
Creatinine (mg/dL | 4 weeks
  Item in comprehensive metabolic panel for safety assessment
Alkaline phosphatase (U/L) | 4 weeks
  Item in comprehensive metabolic panel for safety assessment
Alanine transaminase (ALT) (U/L) | 4 weeks
  Item in comprehensive metabolic panel for safety assessment
Aspartate aminotransferase (AST) (U/L) | 4 weeks
  Item in comprehensive metabolic panel for safety assessment
Calcium (mg/dL) | 4 weeks
  Item in comprehensive metabolic panel for safety assessment
Carbon Dioxide (mmol/L) | 4 weeks
  Item in comprehensive metabolic panel for safety assessment
Chloride (mmol/L) | 4 weeks
  Item in comprehensive metabolic panel for safety assessment
Potassium (mmol/L) | 4 weeks
  Item in comprehensive metabolic panel for safety assessment
Sodium (mmol/L) | 4 weeks
  Item in comprehensive metabolic panel for safety assessment
Total bilirubin (mg/dL) | 4 weeks
  Item in comprehensive metabolic panel for safety assessment
Total protein (g/dL) | 4 weeks
  Item in comprehensive metabolic panel for safety assessment
Body mass index (BMI) | 4 weeks
  Determine whether body mass index is affected by the consumption of the study product.
Blood pressure (mmHg) | 4 weeks
  Determine whether blood pressure is affected by the consumption of the study product.
Heart rate (BPM) | 4 weeks
  Determine whether heart rate is affected by the consumption of the study product.
Waist circumference (cm) | 4 weeks
  Determine whether waist circumference is affected by the consumption of the study product.
White blood cells (x10E3/uL) | 4 weeks
  Item in complete blood count for safety assessment
Red blood cells (x10E6/uL) | 4 weeks
  Item in complete blood count for safety assessment
Hemoglobin (g/dL) | 4 weeks
  Item in complete blood count for safety assessment
Hematocrit (%) | 4 weeks
  Item in complete blood count for safety assessment
Mean corpuscular volume (fL) | 4 weeks
  Item in complete blood count for safety assessment
Mean corpuscular hemoglobin (pg) | 4 weeks
  Item in complete blood count for safety assessment
Mean corpuscular hemoglobin concentration (g/dL) | 4 weeks
  Item in complete blood count for safety assessment
Red cell distribution width (%) | 4 weeks
  Item in complete blood count for safety assessment
Platelets (x10E3/uL) | 4 weeks
  Item in complete blood count for safety assessment
Neutrophils (%) | 4 weeks
  Item in complete blood count for safety assessment
Lymphocytes (%) | 4 weeks
  Item in complete blood count for safety assessment
Monocytes (%) | 4 weeks
  Item in complete blood count for safety assessment
Eosinophils (%) | 4 weeks
  Item in complete blood count for safety assessment
Basophils (%) | 4 weeks
  Item in complete blood count for safety assessment
Neutrophils (Absolute) (x10E3/uL) | 4 weeks
  Item in complete blood count for safety assessment
Lymphocytes (Absolute) (x10E3/uL) | 4 weeks
  Item in complete blood count for safety assessment
Monocytes (Absolute) (x10E3/uL) | 4 weeks
  Item in complete blood count for safety assessment
Eosinophils (Absolute) (x10E3/uL) | 4 weeks
  Item in complete blood count for safety assessment
Basophils (Absolute) (x10E3/uL) | 4 weeks
  Item in complete blood count for safety assessment
Immature granulocytes (%) | 4 weeks
  Item in complete blood count for safety assessment
Immature granulocytes (Absolute) (x10E3/uL) | 4 weeks
  Item in complete blood count for safety assessment
Safety/tolerability | 4 weeks
  This study will monitor the occurrence and frequency of adverse events and safety, both through participant report and blood chemistry/hematology analyses.
Generalized Anxiety Disorder-7 (GAD-7) scale | 4 weeks
  Validated, self-reported scale for the measurement of anxiety severity. The GAD-7 is a 7-item scale with total scores between 0 and 21. Higher scores indicate higher anxiety severity.
Patient Health Questionnaire (PHQ-8) scale | 4 weeks
  Validated, self-reported scale for the measurement of depression severity. The PHQ-8 is an 8-item scale with total scores between 0 and 12. Higher scores indicate higher depression severity.
Leeds Sleep Evaluation Questionnaire (LSEQ) scale | 4 weeks
  Validated, self-reported scale for the measurement of sleep quality. The LSEQ is a 10-item scale. Each item is scored 0 to 100. Higher scores indicate better sleep quality.
Short Form-20 (SF-20) scale | 4 weeks
  Validated, self-reported scale for the assessment of subjective quality of life. The SF-20 is a 20-item scale. Each item is scored 0-100. Higher scores indicate better subjective quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Stevens, PhD, Principal Investigator — doTERRA International
Locations (1):
- doTERRA International, Pleasant Grove, Utah, United States

IPD SHARING:
Plan to Share IPD: No